CLINICAL TRIAL: NCT01298167
Title: Fast Absorbing Gut Suture Versus Cyanoacrylate Tissue Adhesive in the Epidermal Closure of Linear Repairs Following Mohs Micrographic Surgery
Brief Title: Absorbable Suture Versus Tissue Glue to Repair Defects Following Mohs Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1101007845
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Results first posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-10

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Cyanoacrylate; Fast Absorbing Gut; Mohs Surgery; Epidermal closure method
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyanoacrylate Superior/Inferior (Active Comparator): This arm contains data from only the Cyanoacrylate used on superior ½ of wounds & inferior ½ of wounds in randomized patients to determine the impact of Cyanoacrylate tissue glue versus Fast Absorbing Gut suture.
  Interventions: Device: Cyanoacrylate tissue glue versus Fast absorbing gut
- Fast Absorbing Gut Suture Superior/Inferior (Active Comparator): This arm contains data from only the Fast Absorbing Gut Suture used on superior ½ of wounds & inferior ½ of wounds in randomized patients to determine the impact of Cyanoacrylate tissue glue versus Fast absorbing gut suture.
  Interventions: Device: Cyanoacrylate tissue glue versus Fast absorbing gut

INTERVENTIONS:
Device: Cyanoacrylate tissue glue versus Fast absorbing gut — All wounds will be closed using a linear, bilayered closure method, where the buried intradermal absorbing suture (5-0, Polysorb) will be placed along the length of the incision, consistent with standard surgical procedure. Only patients with wounds with a length of 3cm or greater will be enrolled. Each wound will be measured, and the length divided in half. Half of the surgical wound will be randomly selected (by coin toss) for epidermal reapproximation with cyanoacrylate, whereas the other half will be repaired with 6-0 fast absorbing gut suture in standard running fashion.

SUMMARY:
The purpose of the study is to look at which nonpermanent superficial closure method, cyanoacrylate tissue glue or fast absorbing gut suture, leads to a better cosmetic and functional outcome in repairs of facial wounds after Mohs surgery.

DETAILED DESCRIPTION:
Cyanoacrylate is a rapidly polymerizing topical adhesive commonly used as an alternative to traditional sutures. Both cyanoacrylate and fast absorbing gut suture eliminate the need for suture removal which can represent a significant savings in patient and staff time as well as related healthcare resources. Both cyanoacrylate and fast absorbing gut suture are currently routinely used for epidermal closure at Yale following Mohs micrographic surgery. Physician preference currently dictates which epidermal closure method is chosen for a given surgery.

Cyanoacrylate has been reported to decrease trauma to the epidermal edges, minimize suture tract marks in surgical scars, and decrease the risk of inflammatory reaction to suture material. Cyanoacrylate, however, does not allow for wound eversion.

Wound eversion minimizes the risk of a depressed scar from tissue contraction during healing. As with all sutures, fast absorbing gut suture allows for wound eversion which is reported to maximize the likelihood of a good epidermal approximation. On the other hand, fast absorbing gut suture degrades by proteolysis which can result in an inflammatory reaction. Any inflammatory reaction on the skin while healing can affect the final cosmetic outcome (ie. post-inflammatory hyperpigmentation).

A recent article (Tierney 2009), reported that tissue adhesive may not be as effective in achieving optimal cosmesis as fast absorbing gut for defects on the trunk and extremities. However, we would like to study these two methods for the repair of facial wounds, which are in low tension areas as compared to trunk and extremities. Therefore, it is unknown exactly which of these two method is better than the other in epidermal closure of facial wounds follow Mohs micrographic surgery.

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing and able to give informed consent.
* The subject is willing and able to participate in the study as an outpatient and is willing to comply with study requirements.
* The subject is 18 years of age or older.
* The subject has a diagnosis of a non-melanoma skin cancer on the face requiring Mohs micrographic surgery.
* The subjects also has a final wound length of 3cm or greater.
* The subject is able to abide by the protocol of standard postoperative care and is able to attend standard post-operative visits at 3 months after the surgery.

Exclusion Criteria:

* The subject is on systemic immunosuppressants and/or is an organ transplant recipients.
* The subject has reported or suspected hypersensitivity to cyanoacrylate or fast absorbing gut suture.
* The subject has a dermatologic disease in the target site that may interfere with examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Leffell, MD, Principal Investigator — Yale University
Locations (1):
- Yale Dermatologic Surgery, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Kim J, Singh Maan H, Cool AJ, Hanlon AM, Leffell DJ. Fast Absorbing Gut Suture versus Cyanoacrylate Tissue Adhesive in the Epidermal Closure of Linear Repairs Following Mohs Micrographic Surgery. J Clin Aesthet Dermatol. 2015 Feb;8(2):24-9. PMID 25741400

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyanoacrylate Superior ½ of Wound & FAG Inferior ½ of Wound: Patients wounds were divided in half and Cyanoacrylate was utilized for the superior ½ of the wound & Fast Acting Gut Suture was utilized for inferior ½ of wound.
- FAG Superior ½ of Wound & Cyanoacrylate Inferior ½ of Wound: Patients wounds were divided in half and Fast Acting Gut Suture was utilized for the superior ½ of the wound & Cyanoacrylate was utilized for inferior ½ of wound.
Period: Overall Study
Arm/Group | Cyanoacrylate Superior ½ of Wound & FAG Inferior ½ of Wound | FAG Superior ½ of Wound & Cyanoacrylate Inferior ½ of Wound
Started | 6 | 8
Completed | 5 | 8
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyanoacrylate Superior ½ of Wound & FAG Inferior ½ of Wound | FAG Superior ½ of Wound & Cyanoacrylate Inferior ½ of Wound | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: The Visual Analog or Analogue Scale (VAS)* is designed to present to the respondent a rating scale with minimum constraints. Respondents mark the location on the 10-centimeter line corresponding to their feeling. It also gives the maximum opportunity for each respondent to express a personal response style.
  The scale is interpreted as the greater the scale score (as the score approaches 10), the greater the cosmetic and functional outcome of the healed wound.
  * Aitken, R. C. B. (1969). Measurement of feelings using visual analogue scales. Proceedings of the Royal Society of Medicine. 62, 989 - 993
  * Freyd, M. (1923). The graphic rating scale. Journal of Educational Psychology, 43, 83 - 102
  * Hayes, M. H. S. & D. G. Patterson (1921). Experimental development of the graphic rating method. Psychological Bulletin, 18, 98-99
Time Frame: 3 months
Population: Individuals' wounds were divided in half and then treated with both Cyanoacrylate and Fast Absorbing Gut Suture. Individuals were randomized as to which half of the wound (superior or inferior) would be treated by each of the methods.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cyanoacrylate Superior/Inferior: Combined measures of Cyanoacrylate used on both the superior and inferior halves of wounds.
- FAG Superior/Inferior: Combined measures of Fast Absorbing Gut Suture used on both the superior and inferior halves of wounds.
Arm/Group | Cyanoacrylate Superior/Inferior | FAG Superior/Inferior
Number analyzed (Participants) | 13 | 13
units on a scale | 7.47 (0.81) | 7.97 (1.25)

ADVERSE EVENTS:
Arm/Group | Cyanoacrylate Superior ½ of Wound & FAG Inferior ½ of Wound | FAG Superior ½ of Wound & Cyanoacrylate Inferior ½ of Wound
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes